CLINICAL TRIAL: NCT03781557
Title: Effect of Omega-3 in Cognition of Young Healthy Adult
Brief Title: Effects of Omega-3 Fatty Acids Supplement in Cognition of Young Healthy Adults and in Their Reaction Time of Computerized Test After 3 Months of Taking High-concentrated DHA and EPA Fish Softgels
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sulaiman AlRajhi Colleges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SulimanAC-Omega-3
Record Dates: First submitted 2018-12-12; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Cognition; Brain; Neuroscience
Keywords: Omega-3; DHA fatty acids; EPA fatty acids; Cognition; Brain; Healthy Adult; Fish Oil; Human
MeSH Terms: interventions — Docosahexaenoic Acids; Eicosapentaenoic Acid; Fish Oils; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- High-concentrated DHA (Experimental): High-concentrated DHA fish oil softgels
  Interventions: Dietary Supplement: Docosahexaenoic acid
- High-concentrated EPA (Experimental): High-concentrated EPA fish oil softgels
  Interventions: Dietary Supplement: Eicosapentaenoic acid
- Olive Oil (Placebo Comparator): Olive Oil softgels
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid — High-concentrated DHA
  Other Names: MadreLabs, DHA 700 Fish Oil
  Arms: High-concentrated DHA
Dietary Supplement: Eicosapentaenoic acid — High-concentrated EPA
  Other Names: Sports Research, Omega-3 Fish Oil, Triple Strength
  Arms: High-concentrated EPA
Dietary Supplement: Olive oil — Olive Oil softgels
  Arms: Olive Oil

SUMMARY:
In this trial, the investigators are going to investigate the improvement of cognitive brain domains after ingestion of omega 3 products that have high concentrations of DHA, Docosahexaenoic acid, and EPA, Eicosapentaenoic acid, in comparison to control group young healthy adults. The study will assess the improvement by computerized testing by their reaction time before and after the intervention. The researchers will follow the scientific and ethical regulations prevent any harmful effect on recruited subjects.

DETAILED DESCRIPTION:
Research Question :

Research question: Will daily consumption of omega-3 fish oil improve brain cognitive domains?

Study Methodology Research Design:

A placebo-controlled, double-blinded, 3-armed randomized controlled trial.

Population and Sample :

Our target population will be young, healthy adults, educated academic students which are the students of Sulaiman Alrajhi Colleges in Kingdom of Saudi Arabia.

Regarding the sample size, the investigators will put into consideration the confidence level of 95%. Also, the investigators will take into account the size of our population which is the number of students in Sulaiman Al-Rajhi Colleges. In addition to that, the investigators will consider the margin of error to be around 10%. Taking these variables together will give us an estimated sample size of about 66 students which the investigators will reduce to 60 due to financial limitations.

Sampling strategy:

The investigators will recruit the participants from the students of Suliman Alrajhi Colleges by announcing through the emails and by spreading paper announcements in the campus and the housing for volunteering in the research as subjects and the investigators will try to give the participants activity points after coordinating with the students' affairs department. If more than 60 students volunteered for the trial, then the investigators will choose 60 of them based on the exclusion and inclusion criteria and by random sequence generation.

Plan of subjects' recruitment:

The investigators will recruit our subjects from the students of Suliman Al-Rajhi Colleges, both males and females sectors. The sample size will be 60 students in 3 arms (20 control, 20 high doses of Docosahexaenoic acid, DHA, and 20 high doses of Eicosapentaenoic acid, EPA,). The investigators will take the baseline characteristics and do the preliminary cognitive testing using Psytest, (TAP 2.3.1) software. Recruiting the subjects will be according to the exclusion and inclusion criteria mentioned below. After collecting the sample, the investigators will enroll the subjects in the study 6 students a day. So that the investigators will do the preliminary testing and take the baseline characteristics for 6 students at day 1 and then the day after the same group will start taking the intervention (either high dose DHA or high dose EPA or placebo) and another 6 students will be enrolled and so on. Hence day 10 will be the last day of enrollment and the process of enrollment will take 10 days. So, the investigators are going to have ten groups of subjects allocated randomly to the three arms of the study. After 90 days from the date of the enrollment, each group will be assessed, and the post-intervention testing will be carried out. The investigators will take the informed consent from all participant after explaining everything about the study and the potential side effects of supplements, in addition, to take their written agreement after explaining all their inquiries about the study.

Plan of data collectors' recruitment:

The investigators need the data collectors to help to keep an updated information on the subjects and assisting in the process of distributing the pills and their regular intake and also they will ensure quick communication. The investigators will need ten data collectors so that each data collector will supervise a group of six subjects, and these six students will be randomly assigned as mentioned before.

Randomization:

The investigators will do Block randomization in order to have equal numbers in the three arms of the study. Computer-generated random allocation sequences will be used, www.randomizer.org, and when carried out the randomization will help us avoiding selection bias so that no systematic differences exist. Then, the investigators will distribute the subjects in the three arms of the study randomly.

Blinding:

The investigators will make sure that the soft-gels of the DHA group, EPA group, and placebo group will look the same and taste the same so that blinding is not broken and allocation concealment is ensured. The investigators will also try to make the study double blinded.

Supplements and placebo groups:

The investigators will divide randomly the participants to three main groups who will take two softgels of different supplements which are:

1. EPA-high-concentrated fish oil softgels that will provide 1374 mg of EPA and 500 DHA fatty acids per day out of 2500 mg total fat. The chosen product for this concentration is :

   , Sports Research, Omega-3 Fish Oil, Triple Strength, 1250 mg, 180 Softgels,
2. DHA-high-concentrated fish oil softgels that will provide 1400 mg of DHA fatty acids per day out of 2000 mg of total fat. The chosen product for this concentration is :

   , DHA 700 Fish Oil,
3. Olive oil softgels as a placebo that will be totally 2500 mg of fat The chosen product for this is :

   * Healthy Origin, Extra Virgin Olive Oil softgels,

The softgels will be taken every day by oral administration for 60 days and the participants will be instructed and followed by the investigators to take them after the meal and roughly in the same time to unify any possible factor during taking it. The investigators suggest taking it after launch meal immediately. The supplements will be stored in a healthy, cold, and safe environment to guarantee the bioavailability of the products.

The investigators will try to ensure that all supplements capsules have the same out-shape characteristics like color, shape, and size to enhance the double blinding that the investigators put in our research criteria. In addition, the investigators will bring uniformed containers to store the soft-gels and distribute the soft-gels among them to maintain blinding for researchers. That will be the same during distributing the capsules to the participants and it will be in a good-saving uniformed container.

Safety:

Many supplements of omega-3 are US FDA and Saudi FDA approved and can be found in the approved drugs list of each organization). According to the European Food Safety Authority in 2012 , long-term consumption of EPA and DHA supplements at combined doses of up to about 5 g/day, or EPA alone up to 1.8 g/day appear to be safe for the adult population and does not increase the risk of spontaneous bleeding episodes, or affect glucose homeostasis, immune function or lipid peroxidation.

Data collection and communication:

The investigators will distribute a limited amount of softgels every week and check for taking softgels.

Criteria for stopping follow-up and intervention in the subject:

Allergic reaction or exacerbated side effects that cannot be afforded Failure to daily follow-up and compliance to take the supplementation

Medication use :

Autoimmune disease Significant changes in lifestyle throughout the supplementation interval Including a 6.8 kg weight loss

Analysis:

The investigators will analyze the data using the SPSS software program. Descriptive analysis and statistical Drop-outs from the study will be excluded from the analysis, so the analysis type will be, per protocol analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Young Adult (18-25)

Exclusion Criteria:

* Diet rich in fish oil: subjects should not use a diet rich in omega 3 poly-unsaturated fatty acids, that is defined as more than one portion a week or more than 4 portions a month of the following food items
* Salmon Sardines • Flaxseed oil or whole flaxseed Illicit drug use

  • Medications of mental illnesses or that affect brain functions
* Fish Allergy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-05-29 (Estimated)

PRIMARY OUTCOMES:
Attention | 5 minutes
  it will be measured by Psytest (TAP 2.3.1) computerised test to assess the reaction time related to it by milliseconds
Working memory | 5 minutes
  Working memory can be looked at as a system that keeps the information essential for solving difficult dilemmas and processing multi-level tasks or aspects of a situation in order to bring about a final impression.
  it will be measured by Psytest (TAP 2.3.1) computerised test to assess the reaction time related to it by milliseconds.
Sustained attention | 15 minutes
  it will be measured by Psytest (TAP 2.3.1) computerised test to assess the reaction time related to it by milliseconds.
stimulus-reaction incompatibility (Simon effect) | 3 minutes
  Incompatibility occurs in a conflict situation in which divergent stimulus information has to be processed in parallel, thus triggering different reaction tendencies. The Simon and the Stroop effects (in the Colour-Word Interference Test) are classic examples of this effect.
  The present procedure tests the interference tendency in terms of stimulus-reaction incompatibility (Simon effect) . For this test, arrows that are directed to the left or the right are presented on the left or the right of a fixation point. Depending on the direction of the arrow, the test person should respond with the right or left hand irrespective of the side on which the arrow is presented.
Go/ No go | 5 minutes
  this test will measure the specific ability of the subject to suppress an inappropriate response and to react only on the appearance of some stimuli and not in the presence of others, which requires significant central intervention.
  it will be measured by Psytest (TAP 2.3.1) computerised test to assess the reaction time related to it by milliseconds.
Divided attention | 10 minutes
  In this test, an auditory and a visual task must be taken simultaneously, to measure the subject's ability to carry out more than one task at the same time.
  it will be measured by Psytest (TAP 2.3.1) computerised test to assess the reaction time related to it by milliseconds.
Alertness | 5 minutes
  In this test, we will measure the reaction time. Simple reaction time measurements will be done, in which a diamond appears on the screen at random intervals and to which the subject should respond as quickly as possible by pressing a button.
  it will be measured by Psytest (TAP 2.3.1) computerised test to assess the reaction time related to it by milliseconds.